CLINICAL TRIAL: NCT02832024
Title: Clinical Study of Stent Versus Direct Atherectomy Versus Angioplasty to Treat Lower Limb In-stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuanwuH
Record Dates: First submitted 2015-09-14; First posted 2016-07-13 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-05

CONDITIONS: Atherosclerosis; In-stent Arterial Restenosis
Keywords: stents; atherectomy; femoral artery; popliteal artery; In-stent Restenosis
MeSH Terms: conditions — Atherosclerosis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention: Stents (Active Comparator): Stents group
  Interventions: Device: stent
- Intervention: Atherectomy (Active Comparator): Direct Atherectomy group
  Interventions: Device: plaque excision system
- Intervention: Balloon (Active Comparator): Balloon group
  Interventions: Device: Balloon

INTERVENTIONS:
Device: plaque excision system
  Arms: Intervention: Atherectomy
Device: stent
  Arms: Intervention: Stents
Device: Balloon
  Arms: Intervention: Balloon

SUMMARY:
This is a randomized study comparing Stent Versus Direct Atherectomy Versus Angioplasty to Treat Lower Limb In-stent Restenosis (superficial femoral or popliteal artery).

DETAILED DESCRIPTION:
This is a randomized study comparing Stent Versus Direct Atherectomy Versus Angioplasty to Treat Lower Limb In-stent Restenosis (superficial femoral or popliteal artery).

ELIGIBILITY:
Inclusion Criteria:

Provides written informed consent Willing to comply with follow-up evaluations at specified times Has claudication or rest pain due to peripheral arterial In-stent restenosis Disease located within the femoropopliteal artery Patient has a In-stent restenosis lesion(s) with >50% stenosis documented angiographically Patient has symptoms of peripheral arterial disease classified as Rutherford Category 2 or greater.

Exclusion Criteria:

They were excluded if they had one or more of the following: 1. Acute or subacute lower limb ischemia; 2. Severe calcification lesions; 3. Total occlusions lesions more significant than 10 cm or total occlusion lesions with a suspicion of subintimal wire recanalization 4. untreated ipsilateral iliac artery stenosis>70%, or the distal runoff artery <1 root; 5. Previously lower extremity intervention or surgical graft artery bypass; 6. Severe renal insufficiency, creatinine level greater than 2.5 mg/dL; 7. The patient's platelet count is less than 100,000/uL, antiplatelet or anticoagulant contraindications to required medications; 8. Patients with immune system diseases or malignant tumours; 9. ongoing active infection 10. decompensated congestive heart failure or acute coronary syndrome; 11. Unwillingness to return for future follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Primary Patency Rate | 12 months
  Primary patency is defined as no significant reduction of flow detectable by Duplex ultrasound through the index lesion and no further clinically driven target vessel revascularization performed in the interim. Significant reduction of flow is binary restenosis defined as the diameter stenosis >50% with a peak systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success | 1 day
  Technical success is defined as residual stenosis less than 30% by final angiography and/or a flow-limiting dissection.
freedom from clinically-driven TLR | 12 months
  it is defined as freedom from clinically-driven target lesion revascularization
Major Adverse Events | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization, and significant embolic events, which were defined as causing end-organ damage.
Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yongquan G, Lianrui G, Lixing Q, Xuefeng L, Zhu T, Shijun C, Yingfeng W, Jianming G, Jian Z, Zhonggao W. Plaque excision in the management of lower-limb ischemia of atherosclerosis and in-stent restenosis with the SilverHawk atherectomy catheter. Int Angiol. 2013 Aug;32(4):362-7. PMID 23822938